CLINICAL TRIAL: NCT03699527
Title: Medical Cannabis Registry and Pharmacology
Acronym: Med Can Autism
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Zelda Therapeutics (Unknown)
Responsible Party: Sponsor
Other Study IDs: 17-014628
Record Dates: First submitted 2018-09-12; First posted 2018-10-09 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Autism; ASD
Keywords: medical cannabis
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Multiple questionnaires administered — This is an observational trial

SUMMARY:
The overall goals of this research is to describe the 1) natural history of current use and disposition of medical cannabis products including Cannabidiol (CBD) products, being administered to children as standard of care for the treatment of Autism Spectrum Disorder (ASD), 2) understand the pharmacokinetic and pharmacodynamics of medical cannabis products and 3) provide educational feedback on what is learned to families and care providers to provide evidenced based dosing guidance for these products to the pediatric community.

DETAILED DESCRIPTION:
Part 1 of the study will consist of building a patient registry. Eligible patients will be identified and consented for study participation.Parents/legal guardians will be asked the survey related questions from Social Communication Questionnaire (SCQ), personality structure questionnaire (PSQ), Assessment Battery for Children (ABC2), Behavior Rating Inventory of Executive Function (BRIEF2), and the Screen for Child Anxiety Related Disorders (SCARED) (parent version) if appropriate and ASHD5 Rating for either 5-10 year old or 11-17 year old. The description of each survey is below with a link to more information to the ASHD5. All additional questionnaires are already validated by the Institutional Review Board (IRB).

Registry information (as detailed below) will be gathered and entered into the registry.Each subject will be re-contacted approximately every 12 weeks to ask whether medications (cannabis related or other) have changed, efficacy/side effects have changed, or there have been changes in care or medical history. These new data will be recorded in the registry. Subjects may continue in the study for the duration of medical cannabis use, until they remove themselves from the study, or the study closes. All data will remain coded with a Master log of Subject identification numbers (IDs).

Part 2 of the study consists of pharmacokinetic (PK) evaluation of select subjects.

PK sampling of a select formulations will begin subjects are enrolled into the Registry and have consented to PK sampling. . Subjects will have the opportunity to opt in or out of Part 2 upon the initial informed consent process for Part 1.

Part 3 of study related activities will include analysis and summary of the data on approximately a six month basis.

The investigative team will provide study participants with coded summary statistics of medical cannabis products use in the region (either through email, postal mail). This will also be presented at a community-based meeting that all study participants are invited to attend. The study team recognized that participation in a community event will result in loss of de-identification, but also feel that this will occur on a voluntary basis for all study participants.

The study team hypothesizes that the community educational programs will provide study participants an opportunity to connect with others in the community, share concerns, learn from others and allow the development of community-based support systems.

ELIGIBILITY:
Inclusion Criteria

1. Individuals who consume cannabis products in a state which has legalized medical cannabis for the treatment of ASD related symptoms
2. Individuals who have a diagnosis of autism spectrum disorder

Exclusion Criteria

1. Consumption of cannabis products that are not obtained legally
2. Non English speaking individuals
3. Greater than 21 years of age for entry into Part 2 of the study

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Those diagnosed with autism who are under age 21.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Number of children with ASD who use medical cannabis | 5 years
  The primary objective is to create a registry that will describe the natural history and landscape of medical cannabis and CBD use in the pediatric ASD population.
Maximum Cannabinoid concentrations in pediatric patients with ASD | 5 years
  The PK profile of select medical cannabis products in pediatric patients with ASD will be assessed. PK sampling may be performed in the home or at a CHOP site. All Subjects will undergo PK sampling at predetermined times for the determination of cannabinoid concentrations based on the formulation that is being consumed (e.g. If a subject is taking only CBD, Tetrahydrocannabinol (THC) concentrations will not be measured). PK samples will be obtained either using a micro-sampling approach (home or CHOP) or from an indwelling catheter (CHOP site

SECONDARY OUTCOMES:
Number of families who complete the educational program to assess epidemiologic outcomes | 5 years
  Families will be informed of epidemiologic outcomes through an educational program for families that have participated in the research for those families who opt for this component. Although these are not research in nature, they are a direct result of the proposed research and are included in the protocol to demonstrate the study's deliverables.

CONTACTS AND LOCATIONS:
Overall Officials: Athena Zuppa, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No